CLINICAL TRIAL: NCT07289750
Title: The Effect of Alogliptin Combined With Pioglitazone and Metformin Hydrochloride Tablets on Glucose and Lipid Metabolism and Islet Function in Patients With Type 2 Diabetes Mellitus Complicated With Metabolic Dysfunction-associated Fatty Liver Disease.
Brief Title: The Effect of Alogliptin Combined With Actoplus Met on Glucose and Lipid Metabolism and Pancreatic Function in Patients With T2DM Complicated With MAFLD.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-242
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: T2DM; MAFLD
Keywords: T2DM; MAFLD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Drug: combination treatment
- control group (Active Comparator)
  Interventions: Drug: alone treatment

INTERVENTIONS:
Drug: combination treatment — combination of alogliptin and actoplus met
  Arms: experimental group
Drug: alone treatment — actoplus met
  Arms: control group

SUMMARY:
To compare the efficacy and safety of the combination of alogliptin and actoplus met with that of actoplus met alone in improving the glucose and lipid metabolism and pancreatic function in T2DM patients complicated with MAFLD.

ELIGIBILITY:
Inclusion Criteria:

* 1.Meet the T2DM diagnosis criteria of China's Diabetes Prevention and Control Guidelines (2024 Edition) 2.Meet the MAFLD diagnosis criteria of Guideline for the Prevention and Treatment of Metabolic Dysfunction-associated Fatty Liver Disease (Version 2024) 3.HbA1c: 6.5-9.5%，BMI: 19-35 kg/m2。 4.No hypoglycemic drugs or insulin have been used within half a year.

Exclusion Criteria:

* 1.Severe infections, surgeries and other stressful situations. 2.Other types of diabetes. 3.Severe cardiovascular, brain, liver and kidney disorders. 4.Acute complications of diabetes. 5.Malignant tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
hemoglobin A1c | after 6 months of treatment